## Official Title:

Senior PharmAssist: Co-Design and Evaluation of a Toolkit to Promote Scalable Implementation

NCT#: NCT05278650

Informed consent document date: 10/25/2022





Study # Pro00110307

Senior PharmAssist™ Scalability Evaluation Information Sheet

Thank you again for your interest and for agreeing to participate in our pilot **research** project. This **year-long project** aims to evaluate the potential to spread an established program, Senior PharmAssist<sup>TM</sup>, which is designed to improve function and quality of life of older adults with limited incomes, to communities outside of Durham, NC.

With input from community stakeholders interested in implementation of the Senior PharmAssist model, we will work with members of your community to refine and implement existing Senior PharmAssist replication tools. These tools include community readiness assessments, educational tools to facilitate implementation of care processes, and data collection tools for quality improvement.

We are interested in your perspective on the readiness and interest in your community to develop and implement a program to improve health outcomes for older adults with limited incomes. We are specifically interested in efforts to improve medication management and access, tailored community referrals, and Medicare counseling.

We will conduct a series of approximately 10 events over the course of 1 year that will include surveys, interviews, focus groups, co-design workshops, and learning collaborative sessions, conducted over the internet, by phone, or through a videoconferencing platform such as Zoom, and possibly one or two sessions in-person. We plan to audio record the sessions so that we can concentrate on your feedback and ideas rather than taking notes during sessions. Your participation is voluntary and will take no more than 90 minutes per session. You can skip any question or conclude this discussion at any time without any penalty.

The only risk to your participation is the potential for loss of privacy. We will manage that risk by discarding the recordings after data analysis is completed, and by presenting individual answers using a pseudonym (fake name).

We believe you may benefit from having input into designing approaches to implementing a new program that has been shown to improve the wellbeing of older adults with limited incomes who are living in the community.

Only study collaborators at Senior PharmAssist and Duke University and will have access to study information and your responses and identity will be kept confidential. A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. Before we move forward, are there any questions? And do I have your permission to audio-record? We can still proceed if you prefer we don't record at this time.

If you have questions about the research, or your treatment as a research subject, you may call the principal investigator, Dr. Eleanor McConnell at 919-684-9229 or the Duke Institutional Review Board at 919-668-5111.